CLINICAL TRIAL: NCT05064982
Title: The Impact of Paternal Involvement on Breastfeeding
Brief Title: Paternal Involvement in Breastfeeding
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Perran Boran, Professor of Pediatrics, Marmara University
Other Study IDs: 09.2021.845
Record Dates: First submitted 2021-09-16; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Breastfeeding; Paternal Behavior; Depression
Keywords: depression; breastfeeding; paternal depression; paternal involvement; marital relationship
MeSH Terms: conditions — Breast Feeding; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Paternal involvement in breastfeeding has been identified as a significant predictor in maternal breastfeeding outcomes. The main aim of this study is to examine the relationship between reported paternal breastfeeding support and paternal-infant attachment with exclusive breastfeeding and total breastfeeding duration. The hypothesis is that paternal involvement in breastfeeding increase exclusive breastfeeding rates, total breastfeeding duration and strengthen paternal-infant attachment.

DETAILED DESCRIPTION:
Initiation, duration and exclusivity of breastfeeding are greatly influenced by paternal involvement in breastfeeding. Previous studies showed that fathers who are involved in the breastfeeding process have stronger attachments with their babies. However, research on fathers' involvement in their partners' breastfeeding is lacking and there are no comprehensive studies conducted on the effects of the paternal involvement and infant attachment on exclusive breastfeeding (EB) and total breastfeeding duration. Therefore, the aim of the study is to examine the relationship between fathers reported breastfeeding support and paternal-infant attachment with exclusive breastfeeding and total breastfeeding duration. Data will be collected from a tertiary university hospital. The study will be conducted in two phases. In the first phase, the researcher will approach healthy, term, one month old babies and their fathers who fulfilled the eligibility criteria and will invite them to participate in the study. Informed consent will be obtained from participating fathers. The Partner Breastfeeding Influence scale will be used to measure fathers' involvement in their partner's breastfeeding, Paternal-infant attachment, paternal depression, and marital adjustment will be measured with Paternal-Infant Attachment Questionnaire, Edinburgh Postpartum Depression Scale and Marital Adjustment Scale respectively. Four sets of questionnaires will be administered at two time points for the study. The first set will be administered at postpartum first month. The second set of data will be collected at postpartum six months. In the second phase, fathers participating in the study will be interviewed for breastfeeding duration and factors associated with cessation will be explored at postpartum 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

Fathers of

* one-month-old,
* healthy,
* breastfed infants

Exclusion Criteria:

* Infants with a birth weight less than 2500 grams
* Infants who are less than 37 weeks gestation
* Infants with prenatally suspected or diagnosed congenital defects
* Parents with major depression
* Divorced or separated couples

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Fathers
Study Population: Fathers of one-month-old, term, healthy, breastfed infants
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Exclusive breastfeeding duration | at 6 months
  Exclusive breastfeeding duration will be asked with a single question at six months
Total breastfeeding duration | at 12 months
  Total breastfeeding duration will be asked with a single question at 12 months
Total breastfeeding duration | at 24 months
  Total breastfeeding duration will be asked with a single question at 12 months

SECONDARY OUTCOMES:
Change in perceived paternal breastfeeding support | Baseline (postpartum 1st month) and 5 months after (at 6th Month)
  The Partner Breastfeeding Influence Scale (PBIS) will be used to measure perceived breastfeeding support and will be assessed using five dimensions of partner breastfeeding support. These are Savvy, helping, appreciation, breastfeeding presence, and responsiveness. Mean scores are calculated from all questions, from 1 (extremely not supportive) to 5 (extremely supportive) for each breastfeeding support component. High scores show that breastfeeding support of father is notable.
Change in Paternal-Infant Attachment | Baseline (postpartum 1st month) and 5 months after (at 6th Month)
  The Paternal-Infant Attachment Scale (PIAS) will be used to measure the strength of the bond between the father and infant. The PIAS is a scale consisting of 19 items, with every item graded between 1 and 5 points. High scores show that the attachment is strong. The gathered score average from PIAS is near the score of 19 (minimum value) show a weak attachment; however, when it is near the score of 95 (the maximum value), show a strong attachment.
Change in paternal depression | Baseline (postpartum 1st month) and 5 months after (at 6th Month)
  The Edinburgh Postpartum Depression Scale (EPDS) will be used to detect depression as a screening tool. The EPDS is a ten item self-report questionnaire. Items 1 and 2 assess anhedonia; item 3: self-blame; item 4: anxiety; item 5: fear or panic; item 6: inability to cope; item 7: difficulty sleeping; item 8: sadness; item 9: tearfulness and item 10: self-harm ideas. Responses are scored as 0, 1, 2 and 3 according to the increasing severity of the symptoms. Total score is calculated by adding each score of each 10 items. The value of score can range from 0 to 30. The traditional cut-off score for the Edinburgh Postpartum Depression Scale when assessing women is 13 or greater however, a lower cut-off score is recommended for fathers as men express emotions differently from women, mainly that they are less expressive with their negative emotions. For this study a cut-off score of 10 or above will be used to assess Paternal Postpartum Depression.
Change in Marital Adjustment | Baseline (postpartum 1st month) and 5 months after (at 6th Month)
  The Marital Adjustment Scale (MAS) consists of 15 items that evaluate general adjustment, conflict resolution, attachment, and communication. High scores from this scale indicates high marital adjustment. The value of score can range 0 to 60. A score of less than a 43 or below reflects marital distress in marital adjustment scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No